CLINICAL TRIAL: NCT04645095
Title: Which Type of Transcutaneous Electrical Nerve Stimulation is More Effective in Myofascial Pain Syndrome? A Randomized Controlled Trial
Brief Title: Which Type of Transcutaneous Electrical Nerve Stimulation is More Effective in Myofascial Pain Syndrome?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Birkan Sonel Tur, Professor; MD, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-427-16
Record Dates: First submitted 2020-11-23; First posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Myofascial Pain Syndromes
Keywords: Myofascial Pain Syndromes; Transcutaneous Electrical Nerve Stimulation
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional TENS (Active Comparator): Frequency:80 Hz, duration:100 μs
  Interventions: Device: Transcutaneous electrical nerve stimulation; Device: Hot pack
- Burst TENS (Active Comparator): Frequency:100 Hz, fr mod: 0, 200 µs, 2 Bps Hz
  Interventions: Device: Transcutaneous electrical nerve stimulation; Device: Hot pack
- Modulated TENS (Active Comparator): Frequency:80 Hz, fr mod: 50%, Amplitude mode: 40%, duration: 200 µs
  Interventions: Device: Transcutaneous electrical nerve stimulation; Device: Hot pack

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation — All groups were administered hotpack for 20 minutes, different types of TENS therapy for 20 minutes, 5 days a week, total of 15 sessions.
  Other Names: TENS
Device: Hot pack — All groups were administered hotpack for 20 minutes, different types of TENS therapy for 20 minutes, 5 days a week, total of 15 sessions.

SUMMARY:
The aim of this project is to compare the effects of conventional, burst and modulated TENS primarily on pain level, number of trigger points, pressure pain threshold, neck joint range of motion and disability in MAS treatment.

DETAILED DESCRIPTION:
Myofascial pain syndrome (MAS) is a regional pain syndrome characterized by trigger points detected by one or several muscle groups and reflected pain manifestation caused by palpation of these points. Transcutaneous electrical nerve stimulation (TENS) is a physical therapy modality that provides an analgesic effect by delivering a controlled low voltage electrical current to the nervous system through electrodes placed on the skin. Knowledge on how modulation parameters such as frequency, wave width and form alter TENS activity are limited.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of myofascial pain syndrome according to the criteria defined by Travell and Simons

Exclusion Criteria:

* The onset of symptoms is less than 3 months
* Severe cervical disc hernia, radiculopathy or myelopathy
* Stage 3-4 cervical degeneration
* Tumoral, infectious, psychiatric, neurological, uncontrolled systemic disease
* Cardiac pacemaker
* Diagnosed with fibromyalgia syndrome
* Kyphoscoliosis
* Acute trauma history
* Having had previous brain or shoulder surgery
* Injections for MAS and / or physiotherapy programs in the last 3 months
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Measurements will be made before treatment, at the 1st week after treatment and at the 1st month after treatment.
  using Visual Analog Scale score; (0-10); 0 indicates no pain and 10 indicates worst imaginable pain
Number of trigger points in the upper back region | Measurements will be made before treatment, at the 1st week after treatment and at the 1st month after treatment.
  using number
Pressure pain | Measurements will be made before treatment, at the 1st week after treatment and at the 1st month after treatment.
  using algometer (kg/cm2)
Neck joint range of motion | Measurements will be made before treatment, at the 1st week after treatment and at the 1st month after treatment.
  using double inclinometer
Disability | Measurements will be made before treatment, at the 1st week after treatment and at the 1st month after treatment.
  using Modified Neck Disability Index

CONTACTS AND LOCATIONS:
Overall Officials: Birkan Sonel Tur, Prof., Principal Investigator — Ankara University
Locations (1):
- Birkan Sonel Tur, Ankara, Turkey (Türkiye)